CLINICAL TRIAL: NCT03932981
Title: First-line Chemotherapy With Temozolomide Alone for Non-enhancing Adult Brainstem Gliomas, With a Diffuse Subtype and Showing Clinical and/or Radiological Infiltrative Pattern of Progression
Acronym: TEMOTRAD01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160954J; 2018-002654-79 (EudraCT Number)
Record Dates: First submitted 2019-02-04; First posted 2019-05-01 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Adult Brainstem Glioma
Keywords: Brainstem; Adult Glioma; Chemotherapy; Temozolomide
MeSH Terms: conditions — Glioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temozolomide (Experimental): Chemotherapy by temozolomide
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Temozolomide at a monthly standard dose of 150-200 mg/m2/day at day 1 to day 5 for a duration of treatment of 12 months

SUMMARY:
This phase 2 study is a prospective cohort study. Chemotherapy alone will be proposed to adult patients suffering from a "low grade" brainstem glioma subtype showing infiltrative, non-threatening clinico-radiological progression. Patients will receive temozolomide at a monthly standard dose of 150-200 mg/m2/j J1-J5, will be clinically evaluated every month and will undergo radiological evaluation every 2 months. The duration of treatment will be 12 months. Then, the patients will be followed-up until progression, with clinical evaluations and MRI performed every 2-3 months. At the time of recurrence, treatment with focal radiation therapy will be administered (54 Gy in classical fractions).

DETAILED DESCRIPTION:
The goal of this study is to assess the impact (objective response) of first-line chemotherapy in infiltrative non-enhancing adult brainstem gliomas that are progressing in an infiltrative and non-threatening way. Upon progression, (radiotherapy) RT will be administered. Main inclusion criteria are:18 years of age or older/Karnofsky's Index over 50 /Non-enhancing lesion at MRI/Histologically proven infiltrating pattern of brainstem glioma except in case of formal contraindication to surgery determined via discussion of the case with expert neurosurgeons during a national webmeeting ((GLIome du TRonc de l'ADulte group (GLITRAD))/Clinical and/or radiological progression with an infiltrative but non-threatening pattern, warranting antitumoral treatment. The treatment delivered will be Temozolomide at a monthly standard dose of 150-200 mg/m2/day at day 1 to day 5 for a duration of treatment of 12 months. The study is a prospective single-arm phase II trial. Primary end point is objective response rate (radiographic and clinical response) to Temozolomide according to Response assessment in neuro-oncology criteria (RANO criteria). Secondary end points are histological pattern of adult brainstem gliomas/Molecular pattern of adult brainstem gliomas/ Radiological pattern of adult brainstem gliomas based on standard and multimodal MRI/Metabolic pattern of adult brainstem gliomas based on 18F-DOPA PET CT at initial diagnosis and its change after treatment /Global survival/Quality of life questionnaire (EORTC QLQ-C30 with BN-20)/Tolerance to temozolomide/Volumetric velocity of the tumor growth during follow-up before treatment from the initial MRI until the last MRI before beginning of the treatment, established with sagittal cube FLAIR sequences/Volumetric velocity of the tumor growth during follow-up during treatment of chemotherapy, established with sagittal cube FLAIR sequences/Rate of objective response, stabilization and progression under treatment obtained by combining the RANO criteria and the scores obtained on 3 scales (ataxia measured by the Scale for the Assessment and Rating of Ataxia (SARA), diet measured by the Functional Oral Intake Scale (FOIS) and diplopia).A number of 60 patients should be enrolled. THe duration of the study is 4 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Karnofsky's Index over 50
* Non-contrast lesion on MRI
* Histologically proven low grade brainstem glioma with 2 exceptions:

  * formal contraindication to surgery determined via discussion of the case with expert neurosurgeons during a national webmeeting (GLITRAD)
  * negative brainstem biopsy These two exceptions may lead to case-by-case inclusion despite the lack of a histologically-proven diagnosis if clinical and radiological evidence support such a diagnosis and if a very detailed systemic check-up, standardized by the GLITRAD group (spinal MRI, whole body CT, PET, LP (if feasible), blood inflammatory and infectious counts, biopsy of the salivary glands, etc) is negative and allows us to state that this diagnosis is highly probable
* Clinical and/or radiological progression with an infiltrative but non-threatening pattern, warranting antitumoral treatment
* Absolute neutrophil count > 1.5 x 109/l,
* Platelets > 100 x 109/l
* Total bilirubin < 1.5 × ULN,
* AST and ALT< 3 x ULN
* Effective contraception
* Negative pregnancy test (serum beta-HCG) in females of reproductive age
* Written informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Pilocytic astrocytoma
* Ependymoma
* Lack of a histologically proven diagnosis or an uncertain diagnosis regarding the tumoral nature and/or glial nature of the lesion after the GLITRAD webmeeting and a very detailed checkup looking for diagnostic pitfalls
* Contrast enhancement on MRI
* Clinico-radiological data favoring a more aggressive lesion, such as a high grade glioma, even in the case of a "low grade glioma" diagnosis after biopsy, suggesting histological under-grading
* Previous radiotherapy or chemotherapy for this lesion
* Contraindication to Temozolomide (Hypersensitivity to Temozolomide, dacarbazine or severe myelosuppression)
* Contraindication to IRM (pacemaker, intraocular metallic foreign bodies, intracranial metal clips, non-removable hearing aids, neurostimulation electrodes ...)
* Contraindication to IASOdopa® (hypersensitivity)
* Severe renal insufficiency
* Concomitant serious illness unbalanced that may interfere with follow-up
* History of malignancy within 5 years (excluding basal cell carcinoma or in situ carcinoma of the cervix)
* Pregnancy or breastfeeding
* Predictable difficulty with follow-up
* Patient under legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate based on best response (Complete Response (CR) and Partial Response (PR)) to Temozolomide according to RANO criteria. | Baseline, every month for up to 12 months from start of treatment
  A patient will be considered to be in an objective response to Temozolomide if the best response is a complete or partial response defined according to the RANO criteria.

SECONDARY OUTCOMES:
Progression-free survival | 15 months or later, up to 48 months
Histological pattern of adult brainstem gliomas | 15 months
  Description of the histological pattern of adult brainstem gliomas
Molecular pattern of adult brainstem gliomas | 15 months
  Description of the molecular pattern of adult brainstem gliomas
Radiological pattern of adult brainstem gliomas based on standard and multimodal MRI | 15 months
  Description of the radiological pattern of adult brainstem gliomas
Metabolic pattern of adult brainstem gliomas based on 18F-DOPA PET CT at initial diagnosis and its change after treatment | 15 months
  Description of the metabolic pattern of adult brainstem gliomas
Volumetric velocity of the tumor growth before treatment start from the initial MRI until the last MRI before beginning of the treatment, established with sagittal cube FLAIR sequences | Approximatively one month (before beginning of treatment)
  Description of the volumetric growth of adult brainstem gliomas before treatment
Volumetric velocity of the tumor growth during treatment of chemotherapy, established with sagittal cube FLAIR sequences | 12 months
  Description of the volumetric growth of adult brainstem gliomas before treatment
Volumetric velocity of the tumor growth after treatment of chemotherapy, established with sagittal cube FLAIR sequences | up to 48 months
  Description of the volumetric growth of adult brainstem gliomas after treatment
Overall Survival | 15 months or later, up to 48 months
Total score of quality of life measured by European Organization for the Research and Treatment of Cancer Quality of Life questionnaires(EORTC QLQ-C30 and EORTC QLQ-BN20 together) during treatment | Every 2 months up to 12 months
15-month life quality as measured by total score of European Organization for the Research and Treatment of Cancer Quality of Life questionnaires(EORTC QLQ-C30 and EORTC QLQ-BN20 together) | At 15 months
Objective response rate based on best response (CR and PR) to Temozolomide according to RANO criteria combined with total score obtained on three scales (ataxia measured by the SARA scale, diet/swallowing measured by the FOIS scale and diplopia). | Baseline, every month for up to 12 months from start of treatment
  A patient will be considered to be in an objective response to Temozolomide if the best response is a complete or partial response defined according to the RANO criteria and without degradation on the three scales or if the best response is stable according to RANO criteria with an improvement on one on the three scales without degradation of the two others.
  An improvement is defined as an improvement of total score obtained on one of the three scales without degradation of the two others. Stabilization is defined as obtaining the same total score on all three scales. Degradation is defined as degradation of total score on at least one of the scales (even if the score obtained on another scale is improved)
Tolerance to Temozolomide defined by the frequencies and grades of adverse events defined by the CTCAE v5.0 November 27, 2017 | During chemotherapy and until 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence Florence, MD, Principal Investigator — APHP - Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- APHP - Groupe Hospitalier Pitié-Salpêtrière, Paris, France